CLINICAL TRIAL: NCT00753831
Title: Randomized, Double Blind, Active Controlled Study of the Efficacy, Surgical Outcome and Complications of Silicone Rod Sling in Frontalis Sling Suspension Surgery
Brief Title: Efficacy of Aurosling in Frontalis Sling Suspension Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2PR1220827
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Ptosis, Eyelid
Keywords: Blepharoptosis; Ophthalmoplegia; Blepharospasm
MeSH Terms: conditions — Blepharoptosis; Ophthalmoplegia; Blepharospasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Aurosling
  Interventions: Procedure: Aurosling

INTERVENTIONS:
Procedure: Aurosling — Silicon rod to be used in frontalis suspension surgery

SUMMARY:
To Study the Efficacy of Aurosling as a suspension material in Frontalis suspension surgery in ptosis

DETAILED DESCRIPTION:
Silicon rod is an effective and safe material used in frontalis suspension in treating ptosis with poor levator function.The elasticity and ease of adjustment of silicon rod are ideal characteristics for suspension material used to treat severe ptosis in patients with poor bells phenomenon. In the present study , we attend to study the efficacy of aurosling silicon material as a suspension material for frontalis sling surgery

ELIGIBILITY:
Inclusion Criteria:

* Congenital Ptosis
* Severe Ptosis (MRD<0)
* Poor levator function (<4mm by Berke's method)
* Myogenic Ptosis (Myasthenia gravis)
* Chronic progressive external ophthalmoplegia
* Neurogenic Ptosis (Third cranial palsy)
* Blepharospasm
* Ptosis caused by trauma

Exclusion Criteria:

* Acquired Ptosis
* Horners syndrome
* Blepharochalasis/Dermatochalasis
* Mechanical Ptosis
* Mild or Moderate Ptosis (MRD 1>1)
* Good or fair levator function (>4 mm by Berke's method)
* Previous Ptosis surgery
* Ptosis associated syndromes/Other anomalies including
* Marcus Gunn jaw winking syndrome
* Blepharophimosis syndrome
* Dry eye syndromes
* Corneal anesthesia
* Medical/Pediatric/Anesthesia condition contraindicating to surgery or anesthesia
* Nystagmus where adequate measurements could not be done
* Uncorrected vertical squint of any sort

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Ptosis Correction | 15th day, 90th day postoperatively

SECONDARY OUTCOMES:
Adverse Events | 15th day, 90th day postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Usha Kim, DO, Dip NB, Principal Investigator — Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India